CLINICAL TRIAL: NCT02787668
Title: A Carbohydrate-restricted Diet to Reverse Fatty Liver in Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amy Miskimon Goss, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F160218006
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Childhood Obesity; Insulin Resistance
Keywords: childhood obesity; Non-alcoholic fatty liver disease; insulin resistance; carbohydrate-restriction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity; Insulin Resistance | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate-restricted diet (Experimental): This diet is designed to minimize intake of carbohydrate sources such as added sugars, high glycemic grains, and fructose and will provide ≤10% energy from CHO, 25% energy from protein, and ≥65% energy from fat.
  Interventions: Other: Carbohydrate-restricted diet
- Control, low-fat diet (Active Comparator): The control, low-fat diet will contain 55:25:20 %energy from CHO:protein:fat based on the USDA MyPlate Daily Food Plan. For example, an 1800kcal/d plan will include 5 ounces lean meats, 3 cups low-fat dairy, 6 ounces of whole grains, 1 ½ cups fruit, 2 ½ cups vegetables (starchy and non-starchy) and limited fats.
  Interventions: Other: Control, low-fat diet

INTERVENTIONS:
Other: Carbohydrate-restricted diet — Participants will be randomized (20 per group) to the carbohydrate restricted diet (i.e., CHO <10%; fat >65%, protein 25%) or a low fat diet (CHO 55%; fat 20%; protein 25%) for 8 weeks. Individual counseling with the study physician and registered dietitian (RD) will be provided at baseline for initial assessment and diet instruction. Participants will meet with a RD for an individual counselling session at week 2, 4, and 6 of the diet intervention to ensure adherence to the diet prescription. Participants will be encouraged to keep track of dietary intake by using electronic food diaries (weeks 1-8) to review with the RD during individual counseling at week 2, week 4 and week 6.
  Arms: Carbohydrate-restricted diet
Other: Control, low-fat diet — Individual counseling with the study physician and registered dietitian (RD) will be provided at baseline for initial assessment and diet instruction. Participants will meet with a RD for an individual counselling session at week 2, 4, and 6 of the diet intervention to ensure adherence to the diet prescription. Participants will be encouraged to keep track of dietary intake by using electronic food diaries (weeks 1-8) to review with the RD during individual counseling at week 2, week 4 and week 6.
  Arms: Control, low-fat diet

SUMMARY:
The purpose of this study is to determine the effects of a low carbohydrate diet vs a low fat diet on improvement in aminotransferases, hepatic fat infiltration, markers of inflammation, insulin resistance, and body composition in obese adolescents with non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
NAFLD is the most common form of liver disease in children in the United States. Currently, there is no treatment for NAFLD. In adults, weight loss through caloric restriction is commonly recommended to improve fatty liver. Weight loss is particularly difficult for children to achieve and significant caloric restriction may not be a prudent recommendation in developing children and adolescents. Because of this difficulty with weight loss in children, many children go on to develop cirrhosis and eventually undergo liver transplant. Data on the effectiveness of diet to reverse fatty liver and prevent progression to cirrhosis in children is urgently needed. To date, no studies have been done examining how changes in diet composition without intentional caloric restriction influences NAFLD in children. Data from previous studies in adults support the hypothesis that consumption of lower-CHO, higher-fat food sources rich in high-quality proteins and essential fatty acids has beneficial effects on metabolic health in adults without restricting calories. This study aims to test the hypothesis that a low CHO higher- fat diet will induce rapid reversal of fatty liver while also depleting of total and abdominal adiposity, preserving lean mass, and reducing inflammation in adolescents with obesity and NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI over the 85th percentile) male and female adolescents (age range 10-17) with elevated serum aminotransferase levels, diffusely echogenic liver via ultrasound suggestive of fatty liver, and/or prior diagnosis of NAFLD. Participant eligibility will depend on the ability of one parent to attend the initial diet instruction and individual counseling sessions with the registered dietitian during week 2, 4 and 6 of the diet intervention.

Exclusion Criteria:

* Presence of hepatic virus infections (HCV RNA-polymerase chain reaction negative; hepatitis A, B, C, D, E, and G; cytomegalovirus; and Epstein-Barr virus), alcohol consumption, history of parenteral nutrition, and use of drugs known to induce steatosis (for example, valproate, amiodarone, or prednisone) or to affect body weight and carbohydrate metabolism. Autoimmune liver disease, metabolic liver disease, and Wilson's disease will be ruled out by the participants physician prior to enrollment in the study.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in hepatic lipid assessed via magnetic resonance imaging (MRI and magnetic resonance spectroscopy (MRS). | 8 weeks after baseline

SECONDARY OUTCOMES:
Change in body composition via dual-energy X-ray absorptiometry (DXA). | 8 weeks after baseline
Change in liver enzymes via fasting blood draw | At baseline and weeks 2, 4, and 8.
Change in fasting glucose via blood draw | At baseline and weeks 2, 4, and 8.
Change in fasting insulin via blood draw | At baseline and weeks 2, 4, and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Goss, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dowla S, Pendergrass M, Bolding M, Gower B, Fontaine K, Ashraf A, Soleymani T, Morrison S, Goss A. Effectiveness of a carbohydrate restricted diet to treat non-alcoholic fatty liver disease in adolescents with obesity: Trial design and methodology. Contemp Clin Trials. 2018 May;68:95-101. doi: 10.1016/j.cct.2018.03.014. Epub 2018 Mar 27. PMID 29601997